CLINICAL TRIAL: NCT01748851
Title: A Phase III Trial to Evaluate the Efficacy and Safety of the Combination Therapy of Capecitabine and Oxaliplatin (XELOX) in Comparison to the Combination Therapy of Fluorouracil/Folinic Acid and Oxaliplatin (FOLFOX) in Patients With AGC
Brief Title: XELOX Versus FOLFOX for Advanced Gastric Cancer (AGC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor enrollment of patients
Sponsor: Dong-A University Hospital (Other)
Responsible Party: Principal Investigator, Sung Yong Oh, Associate Professor, Dong-A University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCSG ST12-05; ML27924 (Other Grant/Funding Number: Roche Korea Company)
Record Dates: First submitted 2012-12-09; First posted 2012-12-13 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Gastric Carcinoma Stage IV
MeSH Terms: conditions — Stomach Neoplasms | interventions — XELOX; Capecitabine; Folfox protocol; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- XELOX (Experimental): Capecitabine 1000mg/m2 bid D1-D14 Oxaliplatin 130mg/m2 + 5% Dextrose water (5DW) 500ml over 2hour D1 Q 2weeks
  Interventions: Drug: XELOX
- FOLFOX (Active Comparator): Oxaliplatin 85mg/m2 + 5DW 500ml over 2hr D1 Leucovorin 400mg/m2 + 5DW 500ml over 2hr D1 5-Fluorouracil (5-FU) 400mg/m2 IV PUSH D1 5-FU 1200mg/m2 + 5DW 1 Liter over 22hr D1-D2 Q 2weeks
  Interventions: Drug: FOLFOX

INTERVENTIONS:
Drug: XELOX — capecitabine 1000mg/m2 bid po D1-D14
  Other Names: Xeloda
  Arms: XELOX
Drug: FOLFOX — 5-FU 400mg/m2 iv push D1, 5-FU 1200mg/m2 over 22hr D1,D2
  Other Names: 5-FU
  Arms: FOLFOX

SUMMARY:
The purpose of this study is to identify the non-inferiority of the combination therapy of Capecitabine and Oxaliplatin compared with the combination therapy of Fluorouracil/Folinic acid and Oxaliplatin in patients with advanced gastric cancer.

DETAILED DESCRIPTION:
Quality assurance: Data will be collected, controlled, and monitored at the Korean Clinical Study Group (KCSG) data center.

Data will be entered throuGh the E-Case report form (CRF) (Web based data input)

Korean Clinical Study Group (KCSG) data center will do the standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management

Sample size assessment to specify the number of participants or participant years was consulted Statistical specialist. And data analysis will be also discuss with him

Expected median progression-free survival(PFS) in Xelox: 6 months total number of events required: 359 197 patients will be needed After 10% of follow-up loss, 219 patients in each arm, a total of 438 patients will be enrolled

ELIGIBILITY:
Inclusion Criteria:

1. Age :older than 20
2. A patient with at least one measurable primary lesion of which the diameter is confirmed to be 10mm in Spiral CT or multidetector CT (MD CT), or 20 mm or longer in conventional CT (it should be used by a consistent method during the study period). (RECIST v1.1)

   *but, patients who does not have measureable lesion with metastatic resected M1 lymph node or bone metastasis or ascites could be enrolled.
3. No prior palliative chemotherapy (relapse 1 year later after end of adjuvant treatment available)
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 -2
5. The following laboratory test results:

   ① absolute neutrophil count (ANC) ≥1,500/micro Liter (uL), Platelet ≥ 100,000/uL,

   ② aspartate aminotransferase (AST) ≤ 3 x Upper limit of normal (ULN), alanine aminotransferase (ALT) ≤ 3 x ULN , Total bilirubin ≤ 2.0 mg/dL (in case of liver metastasis, 5 x ULN of AST, ALT)

   ③ Creatinine ≤ 1.5 mg/dL
6. A patient who signed the informed consent prior to the participation of the study and who understands that he/she has a right to withdrawal from participation in the study at any time without any disadvantages.

Exclusion Criteria:

1. HER-2 Positive patients
2. Any other malignancies within the past 2 years except curatively treated non-melanoma skin cancer or in situ carcinoma of cervix uteri
3. Subjects who received radiotherapy within 4 weeks prior to randomization
4. Subjects who have chronic or acute infection need to treatment
5. Subjects who received major operation within 4 weeks prior to randomization
6. patients with clinically significant (i.e. active) heart disease (e.g. congestive heart failure, symptomatic coronary artery diseases, cardiac arrhythmias, etc) or myocardial infarction within past 12 months.
7. patient with epilepsy or psychiatric problem including central nervous system(CNS) metastasis.
8. Subjects who not be able to ingestion or have a malabsorption disorder
9. peripheral neuropathy accompany with functional loss
10. Prior history of allergic reaction to study treatment drugs
11. A patient with history of other clinical trial within 4 weeks
12. A patient of childbearing potential without being tested for pregnancy at baseline for positive. (A postmenopausal woman with the amenorrhea period of at least 12 months or longer is considered to have non-childbearing potential.)
13. subject who is decided by investigator decide exclusion with any other reasons

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 6 months after treatment

SECONDARY OUTCOMES:
Response rate | every 6 weeks up to 6 months
overall survival | 3 years later initial study start
performance status (quality of life) | Every 6 weeks up to 1 year
  European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C30 will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Oh, M.D., Principal Investigator — Dong-A University Hospital
Locations (1):
- Dong-A University Hospital, Busan, South Korea